



## **Research Title:**

The Accuracy of Pulp Sensibility Test on Teeth with Deep Periodontal Pocket.

## **Consent Form**

**Date:** 

February 25, 2020





## **Participation Consent Form**

| I | signed below |
|---|---|
| Authorize the doctor to preform the Pulp Sensibility Tests on tooth no. ( lce and electric pulp tester to evaluate the accuracy of pulp sensibility t periodontal pocket. All possible complications have been explained to participation in this study. | est on teeth with dee |
| Signature: | |
| Date: | |